CLINICAL TRIAL: NCT00090142
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, 2-Period, Crossover Study to Evaluate the Effects of a Single Dose of Montelukast on Exercise-Induced Bronchospasm
Brief Title: Montelukast in Exercise-Induced Bronchospasm - 2004 (0476-275)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0476-275; 2004_009
Record Dates: First submitted 2004-08-24; First posted 2004-08-26 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma, Exercise-Induced
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Montelukast - Placebo
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Placebo
- 2 (Experimental): Placebo - Montelukast
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: Montelukast — Montelukast 10 mg tablet administered orally as a single witnessed dose before exercise challenge
Drug: Comparator: Placebo — Placebo tablet administered orally as a single witnessed dose before exercise challenge

SUMMARY:
The purpose of this study is to determine the effect of an approved medication being studied in support of a new approach in the prevention of exercise-induced asthma (a worsening of asthma caused by exercise, also known as exercise-induced bronchospasm), in patients who have a history of worsening asthma after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-to-moderate asthma

Exclusion Criteria:

* Medical history of a lung disorder (other than asthma) or a recent upper respiratory tract infection
* Patient is, other than asthma, not in good, stable health
* The Primary Investigator will evaluate whether there are other reasons why

the patient may not participate

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2004-05; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Philip G, Villaran C, Pearlman DS, Loeys T, Dass SB, Reiss TF. Protection against exercise-induced bronchoconstriction two hours after a single oral dose of montelukast. J Asthma. 2007 Apr;44(3):213-7. doi: 10.1080/02770900701209806. PMID 17454341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized at 8 sites (7 in the US and 1 in Peru).
  Primary therapy period: May to October 2004.
Pre-assignment Details: Patients who required excluded medications, or did not meet FEV1 criteria during the prestudy period were
  excluded from randomization. Patients who required a β-agonist after the exercise challenge and did not
  meet FEV1 criteria within 30 minutes of treatment were also excluded.
Groups:
- Montelukast 10 mg in Period I Then Placebo in Period II: A montelukast 10-mg tablet (Treatment Period I) was taken orally in the
  morning as a single witnessed dose. This was followed by a 3-7 day washout period and then a montelukast
  matching-image placebo tablet (Treatment Period II) was taken orally in the morning as a single witnessed
  dose.
- Placebo in Period I Then Montelukast 10 mg in Period II: A montelukast matching-image placebo tablet (Treatment Period I) was taken
  orally in the morning as a single witnessed dose. This was followed by a 3-7 day washout and then a
  montelukast 10-mg tablet (Treatment Period II) was taken orally in the morning as a single witnessed dose.
Period: Treatment Period I
Arm/Group | Montelukast 10 mg in Period I Then Placebo in Period II | Placebo in Period I Then Montelukast 10 mg in Period II
Started | 31 (1 patient was lost to follow-up after randomization and did not receive any study drug.) | 31
Completed | 26 | 28
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 0 | 1
Period: Treatment Period II
Arm/Group | Montelukast 10 mg in Period I Then Placebo in Period II | Placebo in Period I Then Montelukast 10 mg in Period II
Started | 26 | 28
Completed | 25 | 28
Not Completed | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All randomized patients
Arm/Group | Overall Study Population
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 33
Need for β-agonist rescue medication following exercise challenge [Number; unit: Participants]
  No | 47
  Yes | 15
AUC for percent change from pre-exercise measurement FEV1 in L 0-60 mins after exercise challenge [Mean (Standard Deviation); unit: (percent change) *minutes] — Area under the curve (AUC) for FEV1 percent change from pre-exercise measurement over the first hour after exercise challenge.
  (percent change) *minutes | 815.27 (516.83)
Maximum percent fall in Forced Expiratory Volume in 1 second (FEV1) post-exercise challenge [Mean (Standard Deviation); unit: percent change from pre-exercise measure] — Maximum percent fall in FEV1 from pre-exercise measurement occurring within the first 60 minutes after exercise challenge. Pre-exercise measurement FEV1 is the value [in liters (L)] measured on the day of the exercise challenge, 5 minutes before exercise testing.
  percent change from pre-exercise measure | 26.86 (7.04)
Time to recovery from maximal percent fall [Mean (Standard Deviation); unit: Minutes] — The duration between the time at which the maximum percent fall in FEV1 occurs and the time when FEV1 returns to within 5% of the preexercise baseline for the first time.
  Minutes | 44.73 (32.23)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 2 Hours Post-dose Compared With Pre-exercise Baseline in Patients With Exercise-induced Bronchospasm (EIB)
Description: In patients with EIB, the percent change from pre-exercise baseline FEV, to the lowest FEV1 within 60 minutes after exercise challenge (2 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed 2 hours after a single oral dose
Population: The primary efficacy analysis used the modified intention-to-treat (MITT) approach. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Placebo: All Placebo patients from Treatment Periods I and II
- Montelukast 10 mg: All Montelukast 10 mg patients from Treatment Periods I and II
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 54 | 54
Percent Change | 17.50 (13.82) | 11.70 (10.80)

2. Secondary Outcome: Number of Patients Requiring ß-Agonist Rescue Medication After Exercise Challenge at 2 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 2 hours postdose
Population: The secondary efficacy analysis used a modified
  intention-to-treat (MITT) approach. Patients with data from only one period were not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 54 | 54
Participants
  Patients requiring rescue medication | 7 | 2
  Patients not requiring rescue medication | 47 | 52

3. Secondary Outcome: Number of Patients Requiring ß-Agonist Rescue Medication After Exercise Challenge at 12 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 12 hours postdose
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Participants
  Patients requiring rescue medication | 4 | 2
  Patients not requiring rescue medication | 48 | 50

4. Secondary Outcome: Number of Patients Requiring ß-Agonist Rescue Medication After Exercise Challenge at 24 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 24 hours postdose
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Participants
  Patients requiring rescue medication | 2 | 2
  Patients not requiring rescue medication | 50 | 50

5. Secondary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 12 Hours Postdose Compared With Pre-exercise Baseline in Patients With EIB
Description: In patients with EIB, the percent change from pre-exercise baseline FEV, to the lowest FEV1 within 60 minutes after exercise challenge (12 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed 12 hours after a single oral dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Percent Change | 11.73 (11.64) | 9.87 (11.43)

6. Secondary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 24 Hours Postdose Compared With Pre-exercise Baseline in Patients With EIB
Description: In patients with EIB, the percent change from pre-exercise baseline FEV, to the lowest FEV1 within 60 minutes after exercise challenge (24 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed 24 hours after a single oral dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Percent Change | 10.69 (12.31) | 7.95 (10.80)

7. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60 Min) at 2 Hours Postdose
Description: The measure included only the area below the pre-exercise baseline.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed at 2 hours postdose
Population: The secondary efficacy analysis used a MITT approach. If a patient received β-agonist rescue medication during the 60 minutes following exercise challenge, then the last pre-rescue FEV1 measurement was carried forward to 60 minutes. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: (percent change) *minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 54 | 54
(percent change) *minutes | 582.6 (759.1) | 284.7 (426.9)

8. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60 Min) at 12 Hours Postdose
Description: The measure included only the area below the pre-exercise baseline.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed at 12 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: (percent change) *minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
(percent change) *minutes | 314.0 (417.7) | 241.7 (545.9)

9. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60min) at 24 Hours Postdose
Description: The measure included only the area below the pre-exercise baseline.
Time Frame: Pre-exercise baseline measurement and 0-60 minutes after the exercise challenge performed at 24 hours postdose
Population: The secondary efficacy analysis was an MITT approach. If a patient received β-agonist rescue medication during the 60 minutes following exercise challenge, then the last pre-rescue FEV1 measurement was carried forward to 60 minutes. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: (percent change) *minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
(percent change) *minutes | 269.6 (507.8) | 223.1 (527.1)

10. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 2 Hours Postdose
Description: The time to recovery from maximum percent fall is the duration between the time at which the maximum percent fall in FEV1 after exercise challenge occurs and the time when FEV1 returns to within 5% of the preexercise baseline for the first time.
Time Frame: Exercise challenge at 2 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 54 | 54
Minutes | 34.23 (36.01) | 15.87 (25.29)

11. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 12 Hours Postdose
Description: as for outcome 10
Time Frame: Exercise challenge at 12 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Minutes | 23.40 (32.20) | 9.42 (18.27)

12. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 24 Hours Postdose
Description: as for outcome 10
Time Frame: Exercise challenge at 24 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Montelukast 10 mg
Number analyzed (Participants) | 52 | 52
Minutes | 13.81 (22.80) | 9.47 (19.52)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during Period I and Period II, and up to and including 14 days after the last dose of study therapy
Description: The number of participants listed in the AE table (58 montelukast & 57 placebo) is the number that received treatment.
  Although a participant may have 2 or more AEs they are counted only once in a category. The same participant may appear in other categories.
Arm/Group | Montelukast 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 1/58 | 3/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 10 mg (N=58) | Placebo (N=57)
Headache (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.